CLINICAL TRIAL: NCT02191722
Title: Evaluating the Efficacy of a Comic Book as an Educating Tool for Children With Juvenile Idiopathic Arthritis
Brief Title: "Medikidz Explain JIA Comic Book- Hebrew"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, GIL AMARILYO, MD, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0213-14-RMC
Record Dates: First submitted 2014-07-07; First posted 2014-07-16 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JIA patients (Experimental): All participants will be evaluated before and after reading the comics booklet
  Interventions: Behavioral: reading comics booklet

INTERVENTIONS:
Behavioral: reading comics booklet

SUMMARY:
We believe, that the results of this study will show that children learn from the comic book about their disease, and are now more aware and less frightened about it, and increase their compliance.

DETAILED DESCRIPTION:
We believe, that the results of this study will show that children learn from the comic book about their disease, and are now more aware and less frightened about it, and increase their compliance. If so, it may promote the use of comic books or other fun educational tool in teaching children various other diseases.

ELIGIBILITY:
Inclusion Criteria:

Children with JIA aged 10-18 after parents signed ICF

Exclusion Criteria:

Parents that do not wanf their children to participate in the study.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2014-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
30% or more improvement in a knowledge questionnaire (before and after reading the comics booklet) | 2 Years

SECONDARY OUTCOMES:
10% or higher score in CHQ questionnaire (after reading the comics booklet) | 2 Years
better compliance ( >1 score improvement in 1-5 scale score, as evaluated by the physician after reading the comics booklet). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gil Amarilyo, MD, Principal Investigator — Schneider Children Medical Center of Israel
Locations (1):
- SCMCI, Petah-Tikva, 14 Kaplan S., Israel

REFERENCES:
- [Background] Hampton T. Media lab uses videos, comics, and more to help people understand health issues. JAMA. 2012 Apr 25;307(16):1679-80. doi: 10.1001/jama.2012.507. No abstract available. PMID 22535844